CLINICAL TRIAL: NCT01600612
Title: Oxytocin, Carbetocin and Misopristol for Treatment of Postpartum Hemorrhage: A Multicentric Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Salah M Rasheed, Dr, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: salah-1
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage, oxytocin, carbetocin, misopristol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxytocin (Active Comparator): 30 IU of oxytocin will be given intravenously to patients with atonic postpartum hemorrhage
  Interventions: Drug: oxytocin
- carbetocin (Active Comparator): 10 ug of carbetocin will be given intravenously to patients with atonic postpartum hemorrhage
  Interventions: Drug: carbetocin
- misopristol (Active Comparator): 600 ug of misopristol sublingually will be given intravenously to patients with atonic postpartum hemorrhage
  Interventions: Drug: misopristol

INTERVENTIONS:
Drug: carbetocin — 10 ug of carbetocin will be given intravenously to patients with atonic postpartum hemorrhage
  Other Names: pabal
  Arms: carbetocin
Drug: misopristol — 600 ug of misopristol will be given sublingually to patients with atonic postpartum hemorrhage
  Other Names: Misotac
  Arms: misopristol
Drug: oxytocin — 30 IU of oxytocin will be given intravenously to patients with atonic postpartum hemorrhage
  Arms: Oxytocin

SUMMARY:
Postpartum hemorrhage (PPH) is the leading cause of maternal death worldwide, with an estimated mortality of 140 000 per year. Uterine atony is one of the most important causes of PPH. The traditional treatment of which is the use of uterotonic agents. Oxytocin is the most conventional drug which was proved effective. However, it has the shortcomings of short half life and the necessity of intravenous administration. Misopristol, and more recently Carbetocin were introduced for treatment of atonic PPP not responding to Oxytocin.

Aim of the study is to evaluate the effectiveness of Carbetocin, Misopristol, and Oxytocin for treatment of atonic PPH.

DETAILED DESCRIPTION:
The study will be conducted at the departments of Obstetrics and Gynecology of Sohag, Qena, Al Azhar, and Assuit university hospitals, Egypt. All patients with atonic PPH who delivered vaginally will be invited to participate in the study. Patients who delivered by caesarean section, with retained placenta, with traumatic PPH, associated coagulopathy and those refused to participate in the study will be excluded. The patients will be randomly categorized into 3 groups; the first (n = 100) will receive 30 IU oxytocin intravenously; the second (n = 100) will receive 600 ug misopristol sublingually; the third (n = 100) will receive 100 ug Carbetocin IV. The randomization will be done using opaque sealed envelops containing computer-generated codes. The primary outcome of the study is cessation of bleeding which will be judged by visual inspection of the blood loss by the trialist and by loss of < 300 mL of blood during the first hour after enrollment. The secondary outcomes are time of control of bleeding (minutes), amount of blood loss till control of bleeding (mL), changes in the hemoglobin levels (gm) before and after treatment, Changes in the hematocrite values (%) before and after treatment, the use of additional uterotonic drugs, the rate of complications (%), and the necessity for surgical intervention, and the cost of each medication.

Written consent will be obtained from all participants and approval from the local institutional ethical committee will be included.

ELIGIBILITY:
Inclusion Criteria:

* primary atonic postpartum hemorrhage after vaginal delivery

Exclusion Criteria:

* Patients who delivered by caesarean section
* Retained placenta
* Traumatic postpartum hemorrhage
* Associated coagulopathy
* Chronic medical illness (hepatic , renal diseases)
* Refusal to participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
control of postpartum hemorrhage | within 20 minutes of administration

SECONDARY OUTCOMES:
time of control of bleeding, amount of blood loss till control of bleeding, changes in the hemoglobin and hematocrite levels, use of additional uterotonic drugs, necessity for surgical intervention, and the rate of complications. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Salah M Rasheed, MD, Study Director — Department of Obstetrics and Gynecology, Sohag university, Egypt; magdy M Amin, MD, Study Chair — Department of obstetrics and Gynecology, Sohag university, Egypt; Ahmed H Abd-Ella, MD, Principal Investigator — Department of obstetrics and Gynecology, Qena university, Egypt; Ahmed M Abo Elhassan, MD, Principal Investigator — Department of obstetrics and Gynecology, Assuit university, Egypt; Mazen A El Zahry, M.D., Principal Investigator — Department of Obstetrics and Gynecology, Al Azhar university, Egypt
Locations (1):
- Sohag university, Sohag, Sohag Governorate, Egypt

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518